CLINICAL TRIAL: NCT05301218
Title: CAlcified Lesion Intervention Planning Steered by OCT.
Acronym: CALIPSO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Mutualiste Montsouris (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CARDIO 04 2021
Record Dates: First submitted 2022-03-08; First posted 2022-03-29 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-04

CONDITIONS: Coronary Artery Calcification; Angioplasty
Keywords: Optical Coherence Tomography, OCT; minimal stent area(MSA)
MeSH Terms: conditions — Ornithine Carbamoyltransferase Deficiency Disease | interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- angiography-guided group (Active Comparator): the treatment (including lesion preparation, stent sizing and post implantation optimization) will be performed by angiography. Once the result is considered optimal by the operator, a control OCT run will be acquired.
  Interventions: Procedure: angioplasty
- OCT-guided group (Experimental): a preliminary OCT run will be recorded. An initial predilation with 1.5 to 2.0 mm balloon could be accepted in order to facilitate OCT catheter delivery through the target lesion. The PCI strategy will be guided by a pre-defined algorithm based on initial OCT findings. Post PCI result will be assessed by control OCT and potential optimization steps could be applied according to the results. The MLD-MAX optimization approach will be applied. Final OCT run will be performed at the end of the procedure.
  Interventions: Procedure: angioplasty

INTERVENTIONS:
Procedure: angioplasty — Coronary angioplasty, also called percutaneous coronary intervention, is a procedure used to open clogged heart arteries. Angioplasty uses a tiny balloon catheter that is inserted in a blocked blood vessel to help widen it and improve blood flow to the heart

SUMMARY:
Calcified lesions are very frequent among coronary artery disease stenotic lesions.

The prevalence of calcifications ranges from 30 to 40% (by angiography evaluation) but is higher when analyzed by intra coronary imaging.

Calcified lesions are very frequent among coronary artery disease stenotic lesions. The prevalence of calcifications ranges from 30 to 40% (by angiography evaluation) but is higher when analyzed by intra coronary imaging.

The presence of calcifications increases the risk of adverse evolution after PCI , including stent restenosis, thrombosis and need for repeat revascularisation. Specific and appropriate tools can be used for calcified lesions management , including high pressure non compliant balloons, intravascular lithotripsy and rotablator. Intra vascular OCT has a high sensitivity and specificity for calcium detection among coronary artery lesions. Compared to IVUS, OCT allows a better quantification of calcium sheets (depth extension ) . Several intra coronary imaging based calcified lesions management algorithms have been proposed , but none have been validated in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with chronic coronary syndrome
2. Angiographically moderately to severely calcified target lesion, defined as follows:

   * Moderate: lesion with radio-opacities noted only during the cardiac cycle before contrast dye injection (Aksoy et al., Circ Cardiovasc Interv 2019)
   * Severe: lesion with radio-opacities seen without cardiac motion before contrast dye injection, visible on both sides of the arterial lumen(Aksoy et al., Circ Cardiovasc Interv 2019)
3. Possibility to cross the target lesion with OCT catheter

Exclusion Criteria:

1. On-going cardiogenic shock
2. Acute coronary syndrome related to target lesion
3. Severe renal failure (Creatinine clearance: 30 ml/min/m2)
4. Impossibility to cross target lesion with OCT catheter & balloons,
5. Indication for Rotablator device as first line therapy
6. Pregnancy
7. Age < 18 y
8. Denial to provide consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of the CALIPSO study is the minimal stent area (MSA) on the final OCT run | During the procedure
  The crude minimal stent area (MSA) will be measured along the stent on the target lesion. Stent geometric expansion will be evaluated by the DOCTORS criteria for non-bifurcated segments (Meneveau et, Circulation 2016) and LEMON criteria for bifurcated segments (Amabile et al;, Eurointervention 2020).

SECONDARY OUTCOMES:
Geometrical stent expansion (%) according to the DOCTORS or LEMON criteria | during procedure
  After the stent is deployed, the blood flow dynamics influence the mechanics by compressing and expanding the structure.
Residual post PCI (Percutaneous Coronary Intervention)stenosis (assessed by QCA methods) | during procedure
  Qualitative Comparative Analysis (QCA) is a methodology that enables the analysis of multiple cases in complex situations
Residual major struts malapposition: crude incidence and quantification | during procedure
  malapposition was defined as a lack of contact of at least 1 strut with the underlying vessel wall (at least 150 μm, in the absence of a side branch) with evidence of blood flow behind the strut. It was classified as "major" malapposition if there was evidence of at least 30% of the struts in one frame.
Major adverse cardiovascular events at 30 days and 1 year | at 30 days and 1 year
  Cardiovascular death + Any myocardial infarction + need for re-intervention on the target lesion (TLR)
Peri-procedural MI according to the SCAI definition (23) | during procedure
  according to the SCAI definition (Moussa et al., Journal of the American College of Cardiology 2013)
Coronary artery perforation: incidence | during the procedure and During the full participation period (1 year).]
  Coronary perforation was defined as evidence of extravasation of dye or blood from the coronary artery during or following the interventional procedure
Radiation dose | during procedure
  Differences in dose radiation used during le procedure
Total Contrast medium volume | during procedure
  Differences in amount of contrast drug used during le procedure
Procedure duration | 24th post-operative hour
  differences in duration (time) of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Amabile, MD PhD, Principal Investigator — Institut Mutualiste Montsouris
Locations (14):
- France (14):
  - Ch de Bastia, Bastia
  - CHU de Besançon, Besançon
  - CHU de Bordeaux, Bordeaux
  - Clinique Saint Augustin, Bordeaux
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Louis Pasteur, Le Coudray
  - L'Hôpital Privé du Confluent, Nantes
  - CHU Nîmes, Nîmes
  - Polyclinique les Fleurs, Ollioules
  - CHU de Poitiers, Poitiers
  - Clinique Saint-Hilaire, Rouen
  - Institut Arnaud Tzanck,, Saint-Laurent-du-Var
  - Clinique Pasteur, Toulouse
  - Institut Mutualiste montsouris, Paris, Île-de-France Region

REFERENCES:
- [Derived] Amabile N, Range G, Landolff Q, Bressollette E, Meneveau N, Lattuca B, Levesque S, Boueri Z, Adjedj J, Casassus F, Belfekih A, Veugeois A, Souteyrand G, Honton B. OCT vs Angiography for Guidance of Percutaneous Coronary Intervention of Calcified Lesions: The CALIPSO Randomized Clinical Trial. JAMA Cardiol. 2025 Jul 1;10(7):666-675. doi: 10.1001/jamacardio.2025.0741. PMID 40305015